CLINICAL TRIAL: NCT03103503
Title: Plexa ICD Lead Registry
Status: Terminated | Type: Observational
Why Stopped: Collection of long term lead performance is being transferred to an alternate data collection methodology.
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Plexa Registry
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Results first posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Implantable Defibrillator User

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this registry is to confirm the long-term safety and reliability of BIOTRONIK's Plexa ICD lead.

ELIGIBILITY:
Inclusion Criteria:

* Successfully implanted with a BIOTRONIK ICD or CRT-D compatible system along with the Plexa lead no more than 30 days prior to consent
* Able to understand the nature of the registry and provide informed consent
* Available for follow-up visits on a regular basis at the study site for the expected 5 years of follow-up
* Accepts BIOTRONIK Home Monitoring® concept
* Age greater than or equal to 18 years

Exclusion Criteria:

* Enrolled in any investigational cardiac device trial
* Enrolled in BIOTRONIK's QP ExCELs lead study
* Planned cardiac surgical procedures or interventional measures within the next 6 months
* Expected to receive heart transplantation or ventricular assist device within 1 year
* Life expectancy of less than 1 year
* Patients reporting pregnancy at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject selected for participation should be from the investigator's general patient population according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 901 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Thomas Hospital Research Office, Fairhope, Alabama
  - Jeffrey S Goodman MD, Los Angeles, California
  - Eisenhower Desert Cardiology, Rancho Mirage, California
  - Florida Hospital, Orlando, Florida
  - Advent Health Tampa, Tampa, Florida
  - St. Louis Cardiology Consultants, Alton, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Heartland Cardiology, Wichita, Kansas
  - Research Integrity LLC, Owensboro, Kentucky
  - Northern Light Cardiology, Bangor, Maine
  - University of Michigan, Ann Arbor, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Mercy Clinic Cardiology, Springfield, Missouri
  - St. Louis Heart and Vascular, St Louis, Missouri
  - Gateway Cardiovascular Research Center, St Louis, Missouri
  - Mercy Clinic Heart and Vascular, St Louis, Missouri
  - Glacier View Research Institute Cardiology, Kalispell, Montana
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Novant Health, Winston-Salem, North Carolina
  - Sanford Medical Center, Fargo, North Dakota
  - The Ohio State Wexner Medical Center, Columbus, Ohio
  - Toledo Cardiology, Toledo, Ohio
  - The Arrhythmia Institute, Newtown, Pennsylvania
  - Upstate Cardiology, Greenville, South Carolina
  - Carolina Heart Specialists, Lancaster, South Carolina
  - Carolina Cardiology Associates, Rock Hill, South Carolina
  - Cardiovascular Associates Ltd, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BIOTRONIK Plexa ICD Lead: Subjects consented and implanted with a BIOTRONIK ICD or CRT-D pulse generator and a Plexa lead.
Period: Overall Study
Arm/Group | BIOTRONIK Plexa ICD Lead
Started | 901
Completed | 0
Not Completed | 901
Not completed — Death | 64
Not completed — Physician Decision | 57
Not completed — Withdrawal by Subject | 10
Not completed — Plexa Lead or Pulse Generator Extraction | 10
Not completed — Lost to Follow-up | 3
Not completed — Study Closure | 757

BASELINE CHARACTERISTICS:
Arm/Group | BIOTRONIK Plexa ICD Lead
Number analyzed (Participants) | 901
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data collected and analyzed when available, not all subjects had data available for this measurement.
  years
    number analyzed (Participants) | 894
    (all) | 64.35 (12.59)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data collected and analyzed when available, not all subjects had data available for this measurement.
  Participants
    number analyzed (Participants) | 894
    Female | 237
    Male | 657
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: inches] — Population: Data collected and analyzed when available, not all subjects had data available for this measurement.
  inches
    number analyzed (Participants) | 874
    (all) | 68.5 (4.0)
Weight [Mean (Standard Deviation); unit: pounds] — Population: Data collected and analyzed when available, not all subjects had data available for this measurement.
  pounds
    number analyzed (Participants) | 880
    (all) | 207.2 (57.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Free From Plexa Lead Related Adverse Events
Description: Evaluate the percentage of subjects without an adverse event related to the Plexa lead through study termination. The endpoint is analyzed as the adverse event free-rate. All protocol defined adverse events that occurred more than 30 days after implant and determined to be related to the Plexa lead plus required invasive intervention to resolve or were related to a lead integrity or clinical performance issue were included. Events meeting this criteria but occurring within 30 days were also included except for lead dislodgement, high pacing threshold, failure to capture, or intermittent capture.
Time Frame: Up to 2.5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BIOTRONIK Plexa ICD Lead
Number analyzed (Participants) | 901
percentage of participants | 100.00 [99.49 to 100.00]

2. Secondary Outcome: Plexa Lead Safety-Individual Adverse Events
Description: Evaluate the individual types of adverse events contributing to primary outcome measure 'Percentage of Subjects Free From Plexa Lead Related Adverse Events'
Time Frame: Up to 2.5 years
Population: No primary outcome adverse events were reported; therefore, there are no individual events to be analyzed.
Arm/Group | BIOTRONIK Plexa ICD Lead
Number analyzed (Participants) | 0

3. Secondary Outcome: Pacing Threshold Measurements for the Plexa Lead Through Study Termination
Description: Pacing threshold measurements at pulse width of 0.4 for the Plexa leads at completed follow-up visits.
Time Frame: Up to 2.5 years
Measure: Mean (Standard Deviation); unit: V
Units Other Than Participants: visits with measurement
Arm/Group | BIOTRONIK Plexa ICD Lead
Number analyzed (Participants) | 901
Number analyzed (visits with measurement) | 3714
V | 0.63 (0.28)

4. Secondary Outcome: Sensing Measurements for the Plexa Lead Through Study Termination
Description: Sensing measurements for the Plexa leads at completed follow-up visits.
Time Frame: Up to 2.5 years
Measure: Mean (Standard Deviation); unit: mV
Units Other Than Participants: visits with measurement
Arm/Group | BIOTRONIK Plexa ICD Lead
Number analyzed (Participants) | 901
Number analyzed (visits with measurement) | 3746
mV | 15.88 (5.56)

5. Secondary Outcome: Pacing Impedance Measurements for the Plexa Lead Through Study Termination
Description: Pacing impedance measurements for the Plexa leads at completed follow-up visits.
Time Frame: Up to 2.5 years
Measure: Mean (Standard Deviation); unit: ohms
Units Other Than Participants: visits with measurement
Arm/Group | BIOTRONIK Plexa ICD Lead
Number analyzed (Participants) | 901
Number analyzed (visits with measurement) | 3925
ohms | 567.1 (111.2)

6. Secondary Outcome: Shock Impedance for the Plexa Lead Through Study Termination
Description: Shock impedance measurements for the Plexa leads at completed follow-up visits.
Time Frame: Up to 2.5 years
Measure: Mean (Standard Deviation); unit: ohms
Units Other Than Participants: visits with measurement
Arm/Group | BIOTRONIK Plexa ICD Lead
Number analyzed (Participants) | 901
Number analyzed (visits with measurement) | 3913
ohms | 75.1 (13.7)

7. Secondary Outcome: Percentage of Subjects Free From Protocol Defined Adverse Events
Description: Evaluate the percentage of subjects without a protocol defined and clinical event committee adjudicated adverse event, excluding events included in the primary outcome 'Percentage of Subjects Free From Plexa Lead Related Adverse Events', through study termination. Lead dislodgements, high pacing threshold, failure to capture, and intermittent capture related to the Plexa lead that occurred less than or equal to 30 days after lead implant or a lead revision procedure are included here. The endpoint is analyzed as the adverse event free-rate.
Time Frame: Up to 2.5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BIOTRONIK Plexa ICD Lead
Number analyzed (Participants) | 901
percentage of participants | 95.12 [93.49 to 96.36]

ADVERSE EVENTS:
Time Frame: Though study exit or study termination, an average of 1.1 years
Description: Serious adverse events were defined according to ISO14155.
Arm/Group | BIOTRONIK Plexa ICD Lead
All-Cause Mortality (participants affected / at risk) | 64/901
Serious Adverse Events (participants affected / at risk) | 44/901
Other Adverse Events (participants affected / at risk) | 12/901
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIOTRONIK Plexa ICD Lead (N=901)
Hematoma (Surgical and medical procedures) | 3 (3)
Infection (Infections and infestations) | 11 (11)
Loose set-screw (Surgical and medical procedures) | 3 (3)
Non-healing pocket dehiscence requiring intervention (Surgical and medical procedures) | 1 (1)
Cardiogenic shock during implantation (Surgical and medical procedures) | 1 (1)
Operation wound bleeding (Surgical and medical procedures) | 1 (1)
Venous occlusion associated with the implant procedure (Surgical and medical procedures) | 1 (1)
LV lead related high pacing threshold (Cardiac disorders) | 1 (1)
LV lead related lead dislodgement (Cardiac disorders) | 1 (1)
Twiddler's syndrome (General disorders) | 2 (3)
RV lead related lead dislodgement (Cardiac disorders) | 12 (12)
RV lead related other: high defibrillation threshold.no evidence for lead malfunction (Cardiac disorders) | 1 (1)
RA lead related lead dislodgement (Cardiac disorders) | 5 (6)
Pulmonary Emboli (General disorders) | 1 (1)
RV lead related high pacing threshold (Cardiac disorders) | 1 (1)
RV lead related intermittent capture (Cardiac disorders) | 1 (1)
RV lead related lead impedance out of range, high (Cardiac disorders) | 1 (1)
RV lead related lead undersensing (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIOTRONIK Plexa ICD Lead (N=901)
Hematoma (Surgical and medical procedures) | 2 (2)
Non-healing pocket dehiscence requiring intervention (Surgical and medical procedures) | 1 (1)
Slow wound healing, no sign for infection (Surgical and medical procedures) | 1 (1)
Thrombosis (Surgical and medical procedures) | 1 (1)
LV lead related extracardiac stimulation (Cardiac disorders) | 1 (1)
LV lead related lead impedance out of range, high (Cardiac disorders) | 1 (1)
RV lead related lead dislodgement (Cardiac disorders) | 1 (1)
RV lead related other: positional atrial undersensing (Cardiac disorders) | 1 (1)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1)
RA lead related lead dislodgement (Cardiac disorders) | 1 (1)
RA lead related no capture (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT03103503/Prot_SAP_000.pdf